CLINICAL TRIAL: NCT03554824
Title: Describing Relationships Between Psychosocial Outcomes and Readiness for Transition in Adolescent and Young Adult Patients With Uveitis - a Pilot Study
Brief Title: Psychosocial Outcomes and Transition Readiness in Uveitis
Status: Completed | Type: Observational
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Collaborators: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SCH-2174
Record Dates: First submitted 2018-05-21; First posted 2018-06-13 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pre-Transfer Adolescents aged 10-16 years
- Post-Transfer Young Adults aged 16-25 years
- Parents/Guardians of Pre-Transfer Patients

SUMMARY:
It is widely acknowledged that the transition from paediatric to adult health services should be a multidimensional and multidisciplinary process that addresses the medical, psychosocial, and educational needs of adolescents and young adults (AYA). Despite this, there is currently a scarcity of research examining the relationships between psychosocial factors (e.g., anxiety, social support) and transition readiness in AYA with uveitis. This study therefore aims to examine the relationships between psychosocial factors and transition readiness in pre-transfer adolescents and post-transfer young adults aged 10-25 years diagnosed with JIA at a single centre.

In total, 25 adolescents aged 10-16 years, together with a parent/guardian, will participate at Sheffield Children's Hospital and 10 young adults aged 16-25 years will participate at Sheffield Teaching Hospitals. Participants completed a battery of self-report questionnaire measuring psychosocial factors (anxiety/depression, social support, family functioning, health-related quality of life) and transition readiness (transition knowledge and skills, self-efficacy). Uveitis disease severity was also measured during clinic appointments. A subset of participants will also be asked to take part in a focus group. This study received full ethical approval, and all participants will give their written informed assent or consent before taking part.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of uveitis
* Uveitis managed by either Sheffield Children's NHS Foundation Trust or Sheffield Teaching Hospitals NHS Foundation Trust
* Fluent in English

Exclusion Criteria:

* No diagnosis of uveitis
* Uveitis not managed by either Sheffield Children's NHS Foundation Trust or Sheffield Teaching Hospitals NHS Foundation Trust
* Not fluent in English

Ages: 10 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study population will either be uveitis patients aged 10-25 years or parents/guardians of uveitis patients aged 10-16 years.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
Generalised Anxiety | Day 1, when participants complete the study questionnaire
  Generalised Anxiety Disorder-7 Questionnaire (Spitzer et al., 2006)

SECONDARY OUTCOMES:
Depression | Day 1, when participants complete the study questionnaire
  Patient Health Questionnaire-9 (Spitzer et al., 1999)
Health-related quality of life | Day 1, when participants complete the study questionnaire
  Paediatric Quality of Life Generic Module (Varni et al., 2002)
Social support | Day 1, when participants complete the study questionnaire
  Bath Adolescent Pain Questionnaire Social Support Subscale (Eccleston et al., 2005)
Family functioning | Day 1, when participants complete the study questionnaire
  Bath Adolescent Pain Questionnaire Family Functioning Subscale (Eccleston et al., 2005)
Prosocial and problem behaviours | Day 1, when participants complete the study questionnaire
  Strengths and Difficulties Questionnaire (Goodman, 1997)
Uveitis disease severity | Day 1, during hospital clinic appointment
  Standardization of uveitis nomenclature (SUN) scores will be used to assess uveitis disease severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Children's NHS Foundation Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No